CLINICAL TRIAL: NCT01187745
Title: Evaluation of Twinkling Artifact Compared to Computed Tomography for Evaluation of Kidney Stones
Brief Title: Study to Look for Artifact on Computed Tomography (CT) Representing Kidney Stones
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Dr. Ania Kielar, The Ottawa Hospital
Other Study IDs: 2009520-01H
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Kidney Stones
Keywords: renal calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- suspect kidney stones: Patients presenting with flank abdominal pain
  Interventions: Other: CT Scan followed by ultrasound

INTERVENTIONS:
Other: CT Scan followed by ultrasound — A limited U/S is performed after the CT scan which is ordered by the Emergency Department physician.
  Other Names: CT- computerized tomography; U/S - ultrasound

SUMMARY:
Patients suspected of having a kidney stone are usually evaluated by computed tomography (CT) scan. The investigators hypothesize that ultrasound (U/S) should be sufficient to evaluate kidneys for suspected renal stones.

DETAILED DESCRIPTION:
All patients aged 18 years of age and over who are undergoing a renal stone protocol for evaluation of flank pain will be included.

Pregnant patients will not be included.

ELIGIBILITY:
Inclusion Criteria:

* Adult, able to consent, flank pain

Exclusion Criteria:

* Pregnant, unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with flank pain in the emergency department, suspected to have kidney stones.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The detection of kidney stones on ultrasound compared to CT. | One year

SECONDARY OUTCOMES:
Presence of hydronephrosis, a sign of obstruction of the urinary tract, will also be detected. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ania Kielar, MD FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Civic and General Campuses, Ottawa, Ontario, Canada